CLINICAL TRIAL: NCT03911609
Title: The Influence of Cardiovascular Autonomic Function on Endogenous Pain Modulation Before and After Exercise and Cognitive Task in Fibromyalgia
Brief Title: Cardiovascular Autonomic Function and Endogenous Pain Modulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HR-1812027243
Record Dates: First submitted 2019-04-03; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Fibromyalgia; Exercise; Pain; Autonomic Dysfunction; Physical Activity
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain; Primary Dysautonomias | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All subjects will participate in two randomized sessions (exercise session and cognitive task session). Experimental pain assessment will be performed before after both tasks.
Who Masked: Participant
Masking Description: Participants are masked to the primary hypothesis of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric (Static) Exercise (Experimental): Subjects will perform isometric (static) handgrip exercise at submaximal intensity for four minutes. The exercise will be performed while the subject is seated, and the elbow bent at around 90° and unsupported. Subjects will be asked to rate their pain using numerical pain rating scale that ranges from 0 (no pain) to 10 (worst pain), perceived exertion (RPE) from 0 (Nothing at all) to 10 (extremely strong), and perceived stress from 0 (not stressed at all) to 10 (extremely stressed). The ratings of pain intensity, RPE and perceived stress will be provided before, at the middle and at the end of the exercise.
  Interventions: Other: Exercise
- Cognitive Task (Experimental): The mental math task, which is also known as serial subtraction test, will be performed for four minutes. Subjects will be asked to rate their pain intensity and perceived stress before, at the middle and at the end of the mental math task.
  Interventions: Other: Cognitive Task

INTERVENTIONS:
Other: Exercise — Subjects will perform isometric (static) handgrip exercise at submaximal intensity for four minutes. The exercise will be performed while the subject is seated, and the elbow bent at around 90° and unsupported. Subjects will be asked to rate their pain using numerical pain rating scale that ranges from 0 (no pain) to 10 (worst pain), perceived exertion (RPE) from 0 (Nothing at all) to 10 (extremely strong), and perceived stress from 0 (not stressed at all) to 10 (extremely stressed). The ratings of pain intensity, RPE and perceived stress will be provided before, at the middle and at the end of the exercise.
  Arms: Isometric (Static) Exercise
Other: Cognitive Task — The mental math task, which is also known as serial subtraction test, will be performed for four minutes. Subjects will be asked to rate their pain intensity and perceived stress before, at the middle and at the end of the mental math task.
  Arms: Cognitive Task

SUMMARY:
The study has three aims:

1. To investigate the influence of cardiovascular autonomic function on pain sensitivity at rest in patients with fibromyalgia and age- and sex-matched controls
2. To investigate the influence of cardiovascular autonomic function at baseline and during exercise on the pain response following submaximal isometric exercise
3. To study the relation between the pain response following physical and cognitive tasks (exercise and mental math, respectively).

DETAILED DESCRIPTION:
Fibromyalgia (FM) affects 2 -8% of the population with a higher prevalence in women than men. People with FM report widespread pain that impacts their quality of life. Patients may also experience other symptoms besides pain such as depression, anxiety, fatigue, sleep difficulties and others. Exercise is one of the interventions that have been shown to reduce pain in chronic pain populations. The phenomenon by which exercise reduces pain sensitivity is known as exercise-induced hypoalgesia (EIH). Although exercise is strongly recommended by American Pain Society guideline for the treatment of FM, some patients with FM report an increase in pain and worsening symptoms following acute exercise. The worsening of symptoms may impact adherence to exercise training. Why some people with FM report pain exacerbation while others report pain relief following exercise is not known.

This study aims at assessing the influence of the cardiovascular autonomic nervous system on pain sensitivity at rest and following exercise in patients with fibromyalgia and pain-free individuals.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia
* Healthy Controls without fibromyalgia
* Stable medical management plan for four weeks prior to participation in the study.
* Physical Activity Readiness Questionnaire
* English proficiency

Exclusion Criteria:

* Elbow arthritis
* Carpal tunnel syndrome
* Cardiovascular disease
* Cervical surgery
* Cerebrovascular accident / stroke
* Multiple sclerosis
* Parkinson's disease
* Any central neurodegenerative disease
* Traumatic brain injury
* Peripheral neuropathy of the upper extremity
* Myocardial infarction
* Chronic obstructive pulmonary disease
* Any unstable medical or psychiatric condition
* Diabetes mellitus
* Active cancer
* Lymphedema of the upper extremity
* Claustrophobia
* Raynaud's phenomenon
* Osteoporosis
* Major depressive disorder
* Bipolar disorder
* Rheumatoid arthritis
* Lupus
* Polymyalgia rheumatica
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pressure Pain Threshold to immediately after performance of exercise. | Before and immediately after exercise at session 2 or 3 which is on day 7 or day 21.
  Application of a pressure stimulus to the right forearm and quadriceps muscle at a rate of 50kPa per second until the pressure first becomes painful.
Change from Baseline Pressure Pain Threshold to immediately after cognitive task. | Before and immediately after cognitive task at session 2 or 3 which is on day 7 or day 21.
  Application of a pressure stimulus to the right forearm muscle and quadriceps muscle at a rate of 50kPa per second until the pressure first becomes painful.
Change from Baseline Pressure Pain Threshold to during the submersion of the foot in ice water. | Before and during the submersion of the foot in ice water on session 2 which is day 7 of data collection
  Application of a pressure stimulus to the right forearm muscle and quadriceps muscle at a rate of 50kPa per second until the pressure first becomes painful.
Temporal summation of heat assessment. | the beginning of session 3 which day 21 of data collection
  Subjects will receive ten heat pulses with ramp and return rate of 8˚C/second to the baseline temperature. The peak stimulus interval 0.6 second and the inter-stimulus interval is 0.3 seconds. The baseline temperature will be 39˚C. Subjects will be asked to rate the first, third, fifth, eighth and tenth stimuli.
Heart Rate Variability | baseline, session1 which is day 1 of data collection
  Electrocardiogram data will be recorded for ten minutes. Subjects will be instructed to relax. A two-lead configuration method will be utilized with electrodes placed at right clavicle (negative electrode), left lower rib (positive electrode), and left clavicle (ground electrode).
Change in Heart Rate during Deep Breathing Test | baseline, session 1 which is day 1 of data collection
  The test is done by asking the participant to perform six breathing cycles with each cycle consists of a five seconds inhalation and 5 seconds exhalation (10 second-cycle). Subjects will perform practice trials until they perform respiratory cycles without sudden inhalation or exhalation or holding the breath. Continuous electrocardiogram data will be collected. The change of heart rate during deep breathing test reflects the cardiovascular parasympathetic function. Reduced heart rate variability during deep breathing test indicates reduced parasympathetic tone.
Change in Blood Pressure during Valsalva Maneuver | baseline, session 1 which is day 1 of data collection
  Subjects will be instructed to perform a forceful expiration at a pressure of 40 mm Hg for 15 seconds. This is done by blowing into a syringe that is connected to a pressure gauge, which will be placed in front of the subjects for visual feedback. In addition, feedback of the time will be provided. Continuous blood pressure will be collected during the test. The recovery time of blood pressure to baseline after Valsalva reflects the cardiovascular sympathetic tone. Greater recovery time indicates reduced sympathetic tone.

SECONDARY OUTCOMES:
Total time spent in sedentary and moderate to vigorous physical activity measured by an Actigraph over the course of 7 days. | Worn continuously for a 7-day period during study enrollment.
  An Actigraph is a waist worn device that is used to track the amount and intensity of physical activity performed over the course of seven days. Total time spent in sedentary and moderate to vigorous physical activity is measured in minutes.
Cortisol Awakening Response (CAR) | samples will be collected at home at any day between day 1 and day 7 of data collection
  CAR represents the increase of cortisol levels after awakening particularly in the first 30-45 minutes post-awakening. CAR is normal circadian phenomenon and the increase of cortisol levels post-awakening can range from 50 -150% in healthy adults. CAR can be assessed by taking three samples following awakening (immediately post-awakening, 30 minutes and 45 post-awakening). Reduced CAR indicates a dysfunction in the hypothalamus-pituitary-adrenal axis and reduction in the ability to respond to acute or chronic physiological or psychological stress.
Six-Minute Walk Test | time frame: baseline, day 1 of data collection
  Subjects will be asked to walk as fast as they can on a straight 30 meters walking course for six minutes. The start and end points will be marked with cones. After each minute, subjects will be informed of the time left and standardized encouragement will be provided. Subjects will be asked at the beginning, middle, and end of the test to rate their pain from 0 (no pain) to 10 (worst pain), and to rate their perceived exertion from 0 (nothing at all) to 10 (extremely strong). At the end of the six minutes, subjects will be asked to stop and the distance walked will be measured.
The Fibromyalgia Impact Questionnaire - Revised | on session 1, 2 and 3 which are on day 1,7 and 21 of data collection.
  This questionnaire evaluates the severity of fibromyalgia symptoms over the past 7 days. It has three domains: symptoms, overall impact, and function. The total score ranges from a minimum of 0 to maximum of 210 with higher scores indicating worse function and symptoms.
The Short-Form McGill Pain Questionnaire | on session 1, 2 and 3 which are on day 1,7 and 21 of data collection
  This questionnaire will be used to evaluate the current clinical pain. It evaluates different aspect of pain such as affective, sensory, and cognitive aspects The total score ranges from a minimum of 0 to maximum 45 with higher scores indicating worse symptoms.
Pain Catastrophizing Scale | on session 1 which is day 1 of data collection.
  This is a 13-item scale that evaluates if the subject has an exaggerated negative mental set towards pain. It has 3 sub-scales which are magnification, rumination, and helplessness. Greater scores indicate greater catastrophizing thinking. Rumination scale ranges from 0 to 16 with higher score indicating higher levels of rumination. Magnification scale ranges from 0 to 12 with higher scores indicating higher levels of magnification. Helplessness scale ranges from 0 to 24 with higher scores indicating higher levels of helplessness. The subscale scores are summed to compute a total score ranging from 0 to 52 with higher scores indicating higher levels of pain catastrophizing.
American College of Rheumatology Diagnostic Criteria for Fibromyalgia | Day 1 of data collection
  This questionnaire characterizes the symptoms of those with fibromyalgia. The scale is composed of 3 subscales; widespread pain index, symptom severity score A and B. The widespread pain index ranges from 0 to 19 with 19 indicating greater number of body areas in which pain was experienced. The symptom severity score A ranges from 0 to 9 with 9 indicating greater symptom severity. The symptom severity score B ranges from 0 to 3 with 3 indicating greater number of symptoms experienced. The total Symptom Severity Score is calculated by adding symptom severity score A and symptom severity score B with a total range of 0 (no symptoms) to 12 (great deal of symptoms).
Baseline Lean Mass | 7 days after enrollment.
  Measurement of lean mass with use of dual energy x-ray absorptiometry testing.
Baseline Fat Mass | 7 days after enrollment.
  Measurement of fat mass with use of dual energy x-ray absorptiometry testing.
Composite Autonomic Symptom Score | baseline, session1 which is day 1 of data collection
  This is a 31-item questionnaire that evaluates 6 domains of autonomic nervous system which are secretomotor, orthostatic intolerance, vasomotor, bladder function, gastrointestinal, and pupillomotor. The score ranges from 0 to 100 with higher scores indicating worse autonomic function.
Situational Pain Catastrophizing Scale | in session 2 and 3 which are day 7 and 21 of data collection
  A 6-item questionnaire that explores the negative mental set or catastrophizing thinking in reference to a particular experimental pain experience. The scores ranges from 0 to 24 with higher scores indicating greater situational catastrophizing.
Pain Anxiety Symptom Scale | session 3 which is day 21 of data collection
  This is a 20-item scale that evaluates the pain-related fear or anxiety. It has four domains: cognitive anxiety, avoidance, fearful thinking, and physiological anxiety. The scores range from 0 to 100. The higher the score, the greater the pain-related anxiety.
Depression Anxiety and Stress Scale (DASS21) | session 3 which is day 21 of data collection
  The DASS21 is a questionnaire that evaluates the overall psychological distress. It has three main subscales: depression, anxiety and stress subscale, and each subscale has 7 items. The DASS21 has been validated in chronic pain patients and non-clinical sample. In patients with FM, DASS21 is associated with the severity of symptoms measured with FIQR, and it mediates the relation between pain intensity and disability in patients with chronic low back pain. The scale has three subscales which are depression, anxiety and stress. The score of depression subscale ranges from 0 - 27. The score of anxiety ranges from 0 - 21. The score of stress ranges from 0 - 42. The greater the score in all subscales the worse the outcome.
State Version of State-Trait Anxiety Inventory | on session 1, 2 and 3 which are on day 1,7 and 21 of data collection.
  This is a 20-item questionnaire that evaluates different feelings the subject may or may not have at the moment. The score ranges from 0 to 80 with higher scores indicating greater state anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hoeger Bement, PT, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States